CLINICAL TRIAL: NCT01820156
Title: Diagnosis, Cost and Therapeutic Decision-Making of Home Respiratory Polygraphy for Patients Without High Suspicion of OSA or With Comorbidity - Hospital Polysomnography in Comparison With Three Nights of Home Respiratory Polygraphy
Brief Title: Diagnosis of Patients With Low or Intermediate Suspicion of SAHS or With Comorbidity: Standard Laboratory Polysomnography Compared With Three Nights of Home Respiratory Polygraphy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Jose M. Montserrat, MD PhD. Pulmonary, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 090212TNHRP
Record Dates: First submitted 2013-03-20; First posted 2013-03-28 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2013-09

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- HRP-PSG (Experimental): First performance three nights of HRP and following one night of laboratory PSG
  Interventions: Device: Home Respiratory Polygraphy; Device: Standard Polysomnography
- PSG-HRP (Experimental): First perform laboratory PSG and following three nights of HRP
  Interventions: Device: Home Respiratory Polygraphy; Device: Standard Polysomnography

INTERVENTIONS:
Device: Home Respiratory Polygraphy
Device: Standard Polysomnography

SUMMARY:
Study Objectives: Obstructive sleep apnea (OSA) diagnosis using simplified methods such as home respiratory polygraphy (HRP) is only recommended in patients with a high pre-test probability. The aim is to determine the diagnostic efficacy, therapeutic decision-making and costs of OSA diagnosis using PSG or three consecutive studies of HRP in patients with mild-moderate suspicion of sleep apnea or with co-morbidity that can mask OSA symptoms.

Design and Setting: Randomized, blinded, crossover study of three nights of HRP (3N-HRP) vs. PSG. The diagnostic efficacy was evaluated with ROC curves. Therapeutic decisions to assess concordance between the two different approaches were analyzed by sleep physicians and respiratory physicians (staff and residents) using agreement level and kappa coefficient. The costs of each diagnostic strategy were considered.

DETAILED DESCRIPTION:
Study subjects The study population consisted of subjects who were referred to the sleep unit of the Clínic Hospital, Barcelona, Spain, or the San Pedro de Alcantara Hospital, Cáceres, Spain, with a mild-moderate clinical suspicion of OSA or with notorious co-morbidity that induced frequent symptoms which mimicked those of OSA or could reduce sleep time.

The inclusion criteria were: a) Patients with snoring and/or some observed apneas during sleep. b) Epworth scale less than 15. c) Subjects with notorious co-morbidity. d) Age between 18 and 75 years.

The exclusion criteria were as follows: high suspicion of sleep apnea (heavy snoring, breathing pauses and somnolence that makes social life or working difficult, without any other causes of hypersomnia); diagnosis of OSA; severe heart disease or resistant systemic hypertension; suspicion of non-apneic sleep disorders, such as narcolepsy, REM behavior disorders, and restless leg syndrome; psychophysical disability that would impede the application of the home polygraphy device or major co-morbidity (unstable heart disease, unstable pulmonary disease or disabling stroke); and lack of informed consent for the protocol approved by the ethics committees of the two centres.

Protocol We compared 3N-HRP with laboratory-standard PSG in randomized patients who met the inclusion and exclusion criteria. The subjects were studied on a random basis for one night in a sleep lab (standard PSG) and for three consecutive nights with HRP. Once the first test had started, the second test was scheduled for within the following two days. PSG and HRP were scored separately and the technicians and physicians were blinded to any identifying information about the patients, as well as to any previous results.

Measurements Clinical data: Gender, age, weight, height, body mass index (BMI), waist-hip ratio, neck circumference, systolic and diastolic blood pressure, and alcohol intake measured as ≤ 60 gr/day or > 60 gr/day, and tobacco consumption.

Co-morbidity: Notable cardiovascular, metabolic or lung diseases, as well as diagnosis of insomnia, anxiety, depression, fibromyalgia, chronic fatigue syndrome, or psychiatric treatment.

Symptoms related to OSA: Episodes of nocturnal choking, nocturia, morning headache, or morning tiredness. These data were collected in four degrees of intensity (never, sometimes, frequently, and always). Sleepiness was measured by the Epworth Sleepiness Scale and the American Sleep Disorders Association Sleepiness Scale (ASDA).

Other questionnaires: a) FOSQ (Functional Outcomes of Sleep Questionnaire), which assesses the impact of excessive sleepiness on multiple activities of everyday. b) Euroqol-5D (EQ-5D), which is a standardized instrument for use as a measure of health outcome.

Sleep studies. Standard laboratory PSG (Somté PSG, Compumedics Limited 2006, Abbotsford, Victoria, Australia) was performed according to the technical specifications of the American Academy of Sleep Medicine (AASM). The recorded variables were electroencephalogram (EEG), with derivations F4-M1, C4-M1, and O2-M1; electro-oculogram (EOG); chin electromyogram (EMG); leg electromyogram; electrocardiogram (ECG). Respiratory variables measured by linearized nasal pressure prongs and oronasal thermal flow waveform; respiratory effort signals measured by inductive bands that recorded rib-cage and abdominal movements; oxygen saturation; body position and snoring. A type 3 portable sleep apnea testing was used to perform HRP (Sleep&Go, Bitmed, Sibel S.A. Barcelona, Spain). Recorded variables were: flow measured by linearized nasal pressure prongs, thermal flow, body position, rib-cage and abdominal movements measured by inductive bands, and oxygen saturation. After a detailed explanation of the use of the HRP device (set-up and withdrawal) in the hospital setting, it was taken home and returned by the patient after three home studies.

A valid PSG or HRP had at least 180 recorded minutes. Moreover, a valid HRP had to have at least 3 hours of flow or bands and oximetry measurements for scoring. The periods that were considered as "awake" because of erratic breathing were not considered for scoring. Mean values were obtained for the three nights of HRP. If one study was considered not to be valid, this was removed and the mean values were obtained from the other two nights with HRP. If two studies in the same patient were considered not to be valid, the patient was excluded.

The PSG and HRP were scored manually, separately, and blinded by independent technicians. Sleep staging was performed using the standardized AASM criteria. The respiratory variables obtained from HRP and PSG were scored according to the AASM criteria: apnea defined as a drop in the peak signal excursion of ≈90% from the pre-event baseline with a duration ≥ 10 seconds; and hypopnea defined as a discernible reduction in the amplitude of the airflow signal (≈30% of pre-event baseline) of at least 10 seconds of duration, associated with an arousal and/or ≥ 3% oxygen desaturation from the pre-event baseline. For HRP, hypopnea was defined as a discernible reduction in the amplitude of the airflow signal (≈30% of pre-event baseline) of at least 10 seconds of duration, associated with ≥ 3% oxygen desaturation.

Therapeutic decision-making In addition to the real treatment decision of the physicians from the two sleep units, other 15 reviewers (five sleep medicine specialists; five respiratory physicians; and five respiratory resident physicians who had been trained for at least 3 months in a sleep lab) from other 5 sleep laboratories in Spain, via a website showing clinical data from the patients and data from the sleep studies, take the therapeutic decisions. The reviewers chose one of two options: 1) CPAP treatment; 2) no CPAP treatment/other therapeutic measures. Each patient was presented twice (with PSG or HRP information), blinded and non-consecutively. The criteria for recommending CPAP were an AHI between 5 and 30 with significant symptoms or consequences or an AHI ≥30, taking less into account symptoms or consequences, according to the Spanish Sleep Network guidelines.

Statistics It was estimated that, after accepting an alpha risk of 0.05 and beta risk of 0.2 in a two-sided test, 55 subjects were needed for a minimum difference in AHI of 7.0 units to be recognized as statistically significant. The standard deviation was assumed to be 18. A dropout rate of 5% was anticipated.

Outcomes to be studied and statistical analysis The means of the data obtained from the 3N-HRP were compared with PSG data. Student's t-test and Bland-Altman plots were used to determine the agreement of the AHI measurements obtained by PSG and HRP. ANOVA was used to assess the variability between each of the nights of HRP. The efficacy of the diagnostic test was evaluated using sensitivity and specificity; positive and negative likelihood ratios [LR (+) and LR (-)]; and the percentage of patients with positive and negative diagnosis. The post-test probability of obtaining a true positive when the test was positive or negative was calculated, based on the pre-test probability (prevalence of the disease) and the positive and negative LRs. Receiver operating characteristic (ROC) curves were plotted for the mean of the 3N-HRP with the different polysomnographic AHI cut-off points (≥5, ≥10, ≥15, ≥ 30) for OSA diagnosis to determine the best ROC curve based on area under the curve (AUC) measurements.

Therapeutic decision making The reviewers were grouped as sleep medicine specialists, respiratory medicine physicians and resident physicians. A median of the therapeutic decisions of each group was obtained. Agreement level (100 minus the sum of false positives and negatives) and Cohen's kappa coefficient was used to determine the agreement between therapeutic decisions. All the analyses were developed with the "Statistical Package for Social Sciences" (SPSS, 21.0 for Windows; SPSS Inc., Chicago, IL).

Cost analysis We considered the costs of the each diagnostic strategy in an analysis of two equally effective alternatives.

Test, patient and total costs for PSG and HRP The estimated test costs of PSG and HRP were obtained from the financial department from the two hospitals involved. These costs included the following: personnel involved, equipment depreciation, and fungible material. Patient costs were estimated according to the average costs for each patient of traveling from home to hospital and back by taxi. We considered a round trip to the hospital in the case of PSG and two round trips to pick up and return the HRP device. To estimate the costs per patient, the test and patient costs were divided by the number of patients with a valid recording. To obtain the total costs of PSG and HRP we added up the test and patient costs.

Test, patient and total costs for equal diagnostic efficacy for PSG and HRP For PSG, the test cost for equal diagnostic efficacy was the sum of the test cost and the cost of repeated PSGs due to invalid recordings. For HRP, the test cost for equal diagnostic efficacy was the sum of the test cost and the following: the costs of PSG for patients with invalid HRP recordings; the cost of PSG in patients with indeterminate diagnostic results ("gray zone") and false positive and false negative results. To calculate the patient costs for equal diagnostic efficacy, we also considered the transport costs due to repetitions of tests. To calculate the costs per patient, these costs were divided by the number of patients who completed the trial. Total PSG and HRP costs for equal diagnostic efficacy were obtained by adding up the test and patient costs.

ELIGIBILITY:
Inclusion criteria

* Patients with low or medium suspicion of Sleep Apnea
* Patients with notorious comorbidity
* Age between 18 and 75 years
* Capability to fill in written questionnaires

Exclusion criteria

* Patients with high suspicion of sleep apnea
* Serious heart disease, resistant systemic hypertension, Suspicion of non-apneic sleep disorders, such as narcolepsy, REM behavior disorders and restless leg syndrome.
* Patients with diagnosis of SAHS
* Lack of informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Therapeutic decision based on full PSG or respiratory polygraphy data (3 nights) | Three months
  The investigators want to compare the clinical decision between full PSG (CPAP or NO CPAP)and respiratory polygraphy performed during 3 nights (CPAP or NO CPAP) when there is discrepancy between symptoms and data from respiratory polygraphy.

SECONDARY OUTCOMES:
Apnea and Hypopnea Index (AHI) | 3 months
  AHI obtained from full PSG versus the mean values of the 3 respiratory polygraphy nights
Cost-effectiveness analysis | 3 months
  Cost-effectiveness of the 2 different patients' management methods

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Guerrero A, Embid C, Isetta V, Farre R, Duran-Cantolla J, Parra O, Barbe F, Montserrat JM, Masa JF. Management of sleep apnea without high pretest probability or with comorbidities by three nights of portable sleep monitoring. Sleep. 2014 Aug 1;37(8):1363-73. doi: 10.5665/sleep.3932. PMID 25083017